CLINICAL TRIAL: NCT04036903
Title: D-Lung: An Analytics Platform for Primary Lung Cancer Screening, Diagnosis and Management Based on Deep Learning Technology
Brief Title: D-Lung: An Analytics Platform for Lung Cancer Based on Deep Learning Technology
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Department of Computer Science & Engineering, CUHK (Unknown)
Responsible Party: Principal Investigator, Professor Winnie W.C. Chu, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.306
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer
Keywords: Lung nodules; Deep learning
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: computed tomography — thoracic CT examinations for diagnosis, and/or follow-up.

SUMMARY:
Lung cancer is one of main cause of cancer death in worldwide, characterized of low 5-year survival rate of less than 20%. Pulmonary nodule is considered as the typical imaging manifestation in early stage of lung cancer. The National Lung Screen Trial has demonstrated that the mortality rates could decline greatly, by the utility of low-dose helical computed tomography for screen of pulmonary nodules. Thus, automatic detection, diagnosis and management of pulmonary nodules, play the vital roles in computer-aided lung cancer screening and early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspicious lung nodules.
* Thin-layer thoracic CT and pathology examination have been performed for suspicious lung nodules.

Exclusion Criteria:

* Subjects with accompanied lesions on CT images that may interfere to lung nodules analysis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a single institutional retrospective cohort study of patients within hospitals in Hong Kong, who had undergone thoracic CT for suspicious lung nodules.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
accuracy | 2 years
  proportion of true results(both true positives and true negatives) among whole instances
sensitivity | 2 years
  true positive rate in percentage(%) derived by ROC analysis
specificity | 2 years
  true negative rate in percentage (%) derived by ROC analysis
area under curve (AUC) | 2 years
  area under ROC curve in percentage (%)

SECONDARY OUTCOMES:
average number of false positives per scan (FPs/scan) | 2 years
  FPs/scan in number (N) based on free-response receiver operating characteristic (FROC) analysis
competition performance metric (CPM) | 2 years
  Competitive performance metric (CPM) is a criterion used for CAD system evaluation. Based on FROC paradigm, CPM score is computed as an average sensitivity at seven predefined average false positive rates. CPM score ranges from 0 to 1, with higher CPM score indicating better CAD performance.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No